CLINICAL TRIAL: NCT04593745
Title: Intraocular Pressure in Children With ALL Treated With High Dose Steroids
Brief Title: Intraocular Pressure in Children With Acute Lymphoblastic Leukemia (ALL) Treated With High Dose Steroids
Acronym: ALL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0262-18-RMC
Record Dates: First submitted 2020-04-05; First posted 2020-10-20 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: ALL, Childhood; Steroid-Induced Glaucoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ALL AIEOP-BFM induction (Other): Intraocular pressure messured in children treated with steroids
  Interventions: Device: Intraocular pressure measurment

INTERVENTIONS:
Device: Intraocular pressure measurment — Intraocular pressure measurmentt using iCare devise: TONOPEN

SUMMARY:
Childhood ALL patients are treated with high dose steroids. The study will follow the intraocular pressure of children treated in according to an AIEOP-BFM protocol, during the induction phase that will be compared to the pressure before treatment. Potential risk factors for developing elevated intraocular pressure will be estimated.

DETAILED DESCRIPTION:
Children with ALL in Israel are treating according to the BFM ALL Protocol which contains high dose steroid therapy. One of the known side effects of high dose steroids is Intraocular hypertension, glaucoma, and even irreversible optic nerve injury. Early diagnosis of elevated intraocular pressure (IOP) and early therapeutic interventions might help to prevent future ocular damage.

The purpose of this study is to determine the risk of developing evaluate Intraocular pressure during high dose steroid therapy. If elevated IOP will be common enough, we will try to corelate the risk of elevated IOP with potential risk factors, such as initial IOP, WBC at diagnosis, etc.

Intraocular pressure will be measured by ophthalmologists using iCare devise: TONOPEN during general anesthesia at the day of diagnosis of ALL before steroid therapy initiation, and then after 15 and 33 days. Children with elevated IOP will continue ophthalmologists' follow up and treatment as necessary.

All parents or patients' guardians will sign informed consent for participating in the study.

The study group contains all newly diagnosed children with ALL in Schneider Children Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* ALL diagnosis
* treated with an AIEOP-BFM protocol (including steroids)

Exclusion Criteria:

* Any prior eye condition that can affect intra ocular pressure or its measurement

Ages: 1 Month to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-07-09 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
intra-ocular pressure (IOP) | 15 days of steroid treatment
  Elevated IOP will be defined as pressure >21 mmHg; The risk of developing elevated IOP will be correlated with potential risk factors (T ALL vs. B ALL; WBC at diagnosis; initial IOP at diagnosis etc.)
intra-ocular pressure (IOP) | 1 month of steroid treatment
  Elevated IOP will be defined as pressure >21 mmHg; The risk of developing elevated IOP will be correlated with potential risk factors (T ALL vs. B ALL; WBC at diagnosis; initial IOP at diagnosis etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Shlomi Barzilai Birenboim, Principal Investigator — Schneider Children's Medical Hospital
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No
upon request